CLINICAL TRIAL: NCT00197457
Title: Serum Pepsinogens as an Early Diagnostic Marker of H. Pylori Eradication
Brief Title: Pepsinogens as the Early Marker of H. Pylori Eradication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: pepsinogen2005
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-02-01 (Estimated); Status verified 2001-05

CONDITIONS: H. Pylori Infection; Gastric Ulcer; Duodnal Ulcer
MeSH Terms: conditions — Stomach Ulcer

INTERVENTIONS:
Procedure: serum pepsinogen
Procedure: urea breath test

SUMMARY:
Helicobacter pylori (H. pylori) eradication increases the serum pepsinogen (PG) I/PG II ratio and the percentage change in PG I/PG II ratios was found to be a useful marker of H. pylori eradication (e.g., the PG method). We studied whether the PG method could be an early diagnostic marker of H. pylori eradication even in patients persistently treated with a proton pump inhibitor. Sixty-two H. pylori-positive patients underwent H. pylori-eradication therapy, followed by treatment with a PPI to cure ulcers. Serum levels of PG I and PG II were measured before, at the end of, and at 4 weeks after the eradication therapy. At more than one month after the end of treatments, 13C-urea breath test (UBT) was performed. The cut-off values of percentage changes in PG I/PG II ratios for the diagnosis of eradication of H. pylori were set in proportion to PG I/PG II ratios before eradication in accordance with our previous report. Using the results of UBT as the standard, the percentage change in serum PG I/PG II ratios is useful as an early diagnostic marker for judgment of H. pylori eradication irrespective of PPI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with H. pylori infection

Exclusion Criteria:

* Patients without H. pylori infection

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06

PRIMARY OUTCOMES:
Whether the serum pepsinogen could be an early diagnostic marker of H. pylori eradication even in patients persistently treated with a proton pump inhibitor compared with 13C-urea breath test.

SECONDARY OUTCOMES:
Cost-effectiveness for diagnosis of H. pylori eradication by the serum pepsinogen.

CONTACTS AND LOCATIONS:
Overall Officials: Naohito Shirai, MD., PhD., Study Chair — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan